CLINICAL TRIAL: NCT01331109
Title: A Multicenter, Open-label, 52-Week Extension Study to Evaluate the Safety and Efficacy of Milnacipran in Pediatric Patients With Primary Fibromyalgia
Brief Title: Long-Term Safety and Efficacy Study of Milnacipran in Pediatric Patients With Primary Fibromyalgia
Acronym: MyFi
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Cypress Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLN-MD-29
Record Dates: First submitted 2011-03-31; First posted 2011-04-07 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-07

CONDITIONS: Primary Fibromyalgia
Keywords: Fibromyalgia; Pediatric Fibromyalgia; Adolescent Fibromyalgia; milnacipran; Savella; loss of therapeutic response; Forest Research Institute; Pain; Fatigue; Serotonin Norepinephrine Reuptake Inhibitors
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Milnacipran (Experimental): oral administration, twice daily dosing
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Milnacipran — maximum tolerated dose (50, 75, or 100 mg/day tablets); for 52 weeks.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of milnacipran in pediatric patients aged 13 to 17 years with primary fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed or discontinued prematurely from lead-in study, MLN-MD-14, tolerating a minimum daily dose of 50mg milnacipran

Exclusion Criteria:

* Can not tolerate a minimum daily dose of 50mg milnacipran
* Significant risk of suicidality
* Pregnant or breastfeeding

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M D'Astoli, LPN, Study Director — Forest Laboratories
Locations (31):
- United States (31):
  - Forest Investigative Site 040, Birmingham, Alabama
  - Forest Investigative Site 033, Bullhead City, Arizona
  - Forest Investigative Site 012, Fresno, California
  - Forest Investigative Site 045, Fresno, California
  - Forest Investigative Site 051, Fresno, California
  - Forest Investigative Site 035, Orange, California
  - Forest Investigative Site 053, Orange, California
  - Forest Investigative Site 050, Sacramento, California
  - Forest Investigative Site 034, Colorado Springs, Colorado
  - Forest Investigative Site 014, Spring Hill, Florida
  - Forest Investigative Site 055, West Palm Beach, Florida
  - Forest Investigative Site 058, Blue Ridge, Georgia
  - Forest Investigative Site 010, Peoria, Illinois
  - Forest Investigative Site 017, Louisville, Kentucky
  - Forest Investigative Site 009, Ann Arbor, Michigan
  - Forest Investigative Site 024, Rochester Hills, Michigan
  - Forest Investigative Site 036, Stevensville, Michigan
  - Forest Investigative Site 049, Whitehouse Station, New Jersey
  - Forest Investigative Site 018, Albuquerque, New Mexico
  - Forest Investigative Site 062, Raleigh, North Carolina
  - Forest Investigative Site 052, Winston-Salem, North Carolina
  - Forest Investigative Site 016, Cincinnati, Ohio
  - Forest Investigative Site 015, Dayton, Ohio
  - Forest Investigative Site 046, Greer, South Carolina
  - Forest Investigative Site 023, Austin, Texas
  - Forest Investigative Site 003, San Antonio, Texas
  - Forest Investigative Site 042, San Antonio, Texas
  - Forest Investigative Site 025, Clinton, Utah
  - Forest Investigative Site 013, Salt Lake City, Utah
  - Forest Investigative Site 063, Seattle, Washington
  - Forest Investigative Site 004, Racine, Wisconsin

REFERENCES:
- [Derived] Arnold LM, Bateman L, Palmer RH, Lin Y. Preliminary experience using milnacipran in patients with juvenile fibromyalgia: lessons from a clinical trial program. Pediatr Rheumatol Online J. 2015 Jun 26;13:27. doi: 10.1186/s12969-015-0025-9. PMID 26112278

RESULTS

PARTICIPANT FLOW:
Groups:
- Milnacipran: oral administration, twice daily dosing
  Milnacipran : maximum tolerated dose (50, 75, or 100 mg/day tablets); for 52 weeks.
Period: Overall Study
Arm/Group | Milnacipran
Started | 57
Completed | 0
Not Completed | 57
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 1
Not completed — Study Terminated by Sponsor | 38

BASELINE CHARACTERISTICS:
Population: All demographic data was based on the safety population, which consists of 57 patients who took at least 1 dose of open-label milnacipran.
Arm/Group | Milnacipran
Number analyzed (Participants) | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.35)
Age, Customized [Number; unit: participants]
  13 years old | 5
  14 years old | 12
  15 years old | 11
  16 years old | 12
  17 years old | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 57
Maximum Tolerated Dose of Milnacipran [Number; unit: participants] — Maximum tolerated daily dose of milnacipran.
  participants
    Less than 50mg | 0
    50 mg | 3
    75 mg | 8
    100mg | 46

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Number of Patients Who Experienced Level 5 Suicidal Ideation, as Assessed by the Electronic Columbia-Suicide Severity Rating Scale (eC-SSRS).
Description: The electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) is a validated, self-rated version of the C-SSRS designed to uniquely assess both suicidal behavior and ideation. Suicidal ideation is assessed at 5 distinct levels of increasing severity:
  * Level 1: Wish to be Dead
  * Level 2: Non-Specific Active Suicidal Thoughts
  * Level 3: Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act
  * Level 4: Active Suicidal Ideation with Some Intent to Act, without Specific Plan
  * Level 5: Active Suicidal Ideation with Specific Plan and Intent
Time Frame: Baseline (Visit 1) to Week 53 (Visit 9)
Population: 57 patients who took at least 1 dose of open-label milnacipran were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Milnacipran
Number analyzed (Participants) | 57
participants | 0

2. Other Pre Specified Outcome: Number of Patients Who Experienced Level 4 Suicidal Ideation, as Assessed by the Electronic Columbia-Suicide Severity Rating Scale (eC-SSRS).
Description: as for outcome 1
Time Frame: Baseline (Visit 1) to Week 53 (Visit 9)
Population: 57 patients who took at least 1 dose of open-label milnacipran were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Milnacipran
Number analyzed (Participants) | 57
participants | 1

3. Primary Outcome: Adverse Events
Description: Number of Patients who experience one or more treatment emergent adverse event (TEAE)
Time Frame: Baseline (Visit 1) to Week 53 (Visit 9)
Population: 57 patients who took at least 1 dose of open-label milnacipran were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Milnacipran
Number analyzed (Participants) | 57
participants | 42

4. Other Pre Specified Outcome: Number of Patients Who Experienced Level 3 Suicidal Ideation, as Assessed by the Electronic Columbia-Suicide Severity Rating Scale (eC-SSRS).
Description: as for outcome 1
Time Frame: Baseline (Visit 1) to Week 53 (Visit 9)
Population: 57 patients who took at least 1 dose of open-label milnacipran were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Milnacipran
Number analyzed (Participants) | 57
participants | 1

5. Other Pre Specified Outcome: Number of Patients Who Experienced Level 2 Suicidal Ideation, as Assessed by the Electronic Columbia-Suicide Severity Rating Scale (eC-SSRS).
Description: as for outcome 1
Time Frame: Baseline (Visit 1) to Week 53 (Visit 9)
Population: 57 patients who took at least 1 dose of open-label milnacipran were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Milnacipran
Number analyzed (Participants) | 57
participants | 0

6. Other Pre Specified Outcome: Number of Patients Who Experienced Level 1 Suicidal Ideation, as Assessed by the Electronic Columbia-Suicide Severity Rating Scale (eC-SSRS).
Description: as for outcome 1
Time Frame: Baseline (Visit 1) to Week 53 (Visit 9)
Population: 57 patients who took at least 1 dose of open-label milnacipran were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Milnacipran
Number analyzed (Participants) | 57
participants | 3

7. Other Pre Specified Outcome: Number of Patients Who Experienced Any Suicidal Behavior as Assessed by the Electronic Columbia-Suicide Severity Rating Scale (eC-SSRS)
Description: The electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) is a validated, self-rated version of the C-SSRS designed to uniquely assess both suicidal behavior and ideation. Suicidal behaviors as defined by the eC-SSRS are:
  * Preparatory acts or behavior
  * Aborted attempt
  * Interrupted attempt
  * Actual attempt
  * Completed suicide attempt
Time Frame: Baseline (Visit 1) to Week 53 (Visit 9)
Population: 57 patients who took at least 1 dose of open-label milnacipran were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Milnacipran
Number analyzed (Participants) | 57
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected during a 14-month period from July, 2011 to August, 2012.
Arm/Group | Milnacipran
Serious Adverse Events (participants affected / at risk) | 2/57
Other Adverse Events (participants affected / at risk) | 28/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran (N=57)
Cholecystitis (Hepatobiliary disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran (N=57)
Nausea (Gastrointestinal disorders) | 10
Decreased appetite (Metabolism and nutrition disorders) | 6
Tachycardia (Cardiac disorders) | 6
Urinary tract infection (Infections and infestations) | 5
Vomiting (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 4
Heart rate increased (Investigations) | 4
Dizziness (Nervous system disorders) | 3
Hepatic enzyme increased (Investigations) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Weight decreased (Investigations) | 3
Weight increased (Investigations) | 3

LIMITATIONS AND CAVEATS:
This study was terminated early, resulting in a small number of patients analyzed. Only descriptive statistics were presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.